CLINICAL TRIAL: NCT07264218
Title: Clinical Effectiveness of a Patient-tailored Orthosis Based on 3-dimensional (3D) Scanner Modeling and 3D Printing Technology for Microstomia Caused by Burns : Pilot Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Hangang Sacred Heart Hospital, Hangang Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-21
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Burn; 3D Printing; Microstomia; Split Thickness Skin Graft
Keywords: microstomia; mouth; split thickness skin graft; burn; 3D scanner modeling
MeSH Terms: conditions — Burns; Microstomia

STUDY DESIGN:
Intervention Model Description: Manufacturing patient-tailored mouthpiece using 3D modeling technology. The participant was advised to wear the appliance throughout the day except during meals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The participant was advised to wear the appliance throughout the day . (Experimental): The participant was advised to wear the appliance throughout the day
  Interventions: Other: patient's tailored mouthpiece fitting

INTERVENTIONS:
Other: patient's tailored mouthpiece fitting — Manufacturing patient-tailored mouthpiece using 3D modeling technology. The participant was advised to wear the appliance throughout the day except during meals. The maximaum horizontal and vertical distances were measured every two weeks to assess whether the mouthpiece had the ability to stretch against the scar. If the patient found it easy to wear or there was no stretching effect, the patient-tailored mouthpiece was remade.

SUMMARY:
Mircostomia is not clearly defined in terms of size, but is diagnosed when it causes difficulty in eating, pronounciation, or maintaining oral hygiene. Although various treatments have been applied to microstomia caused by mouth contracture after facial burns, there is no established protocol yet. This study aimed to confirm the clinical usefulness of patient-customized mouthpiece using 3D scanner modeling and printing technology.Each participant's mouths were scanned using a 3D scanner (Peel 3, Peel 3D, Canada). The scanned model was imported into the modeling software (Geomagic Design X, 3D Systems, USA). After modeling the mouthpiece to fit the maximum horizontal and vertical length of the mouth and the thickness of the lips, it was manufactured using a 3D printer (Form 4B Medical, Formlabs, USA). The participant was advised to wear the appliance throughout the day except during meals. As a primary outcome, the vertical and horizontal distances of the mouth were measured before and after wearing the patient-customized mouthpiece for 2 months. As secondary outcomes, the biological scar properties, the Vancouver Scar Scale (VSS), and the Patient and Observer Scar Assessment Scale (POSAS) scores were evaluated.

DETAILED DESCRIPTION:
Introduction Microstomia is defined as a mouth size that becomes so small that it interferes with oral functions such as oral hygiene care, eating, and speaking with oral function after trauma, facial burns, or surgical procedures for skin cancer, although the exact definition is ambiguous due to cultural differences and standards in each country. Therfore, the diagnosis is defined by functional decline and patient-reported discomfort (1). The cause of microstomia are divided into intraoral and perioral causes. Damage to the sphincter action of the orbicularis oris muscles due to perioral causes, such as burns or trauma, causes contracture which limits lip movement when eating or specking. In the cases of burns around the mouth, the degree of functional impairment varies depending on the extent and depth of the scar. Hypertrophic scars occur in deep second burns or more, and the scar increases as it undergoes the inflammatory, proliferative, and remodeling stages of scar healing. Scar formation increases for several months after burn injury, causing abnormal movement of the surrounding tissue and the scar sites (2). There are various causes of microtomia and various symptoms depending on the severity of the damage, so various attempts are being made to improve the symptoms (3). Conservative treatment generally includes physical therapy and massage to improve facial muscle movement and the use of orthosis to prevent the progression of microstomia. To prevent the progression of microstomia during the healing process of scars after trauma or burns, it is recommended to apply a brace within 10 to 14 days after the injury, but ready-made orthosises are difficult to apply to mouth that are too small, children, or those with severe deformities. The creating of a mouthpiece applied to patient with microstomia in the acute phase is a challenging task tha must be realized to improve clinical outcomes.

Optical three-dimensional (3D) scanning and 3D printing are being used for medical applications such as accurate visualization, precise preoperative anatomical measurements, and patient-specific guides (4). These technologies can be used to manufacture patient-specific orthosis for preventing post burn contractures (5). The technologies have the advantage of saving time and cost in the production of personalized devices and of being able to accurately measure the paricipant's body (6, 7). 3D scanning and printing technology is used for patient-specific body measurements on curved body parts such as the face, hands, and neck, which are difficult to apply with ready-made orthosis (5, 6, 8, 9). The ideal personalized 3D orthosis wound be created by scanning to get the most realistic and accurate outline of the body (10).

There has been little research on the use of 3D scanning modeling technology to produce mouthpiece for patients with microstomia caused by surgery including split thickness skin grafting after burns or cancer operations. This study aimed to confirm the clinical effectiveness of applying patient-tailored mouthpiece using 3D scanning and 3D printing technology to microstomia caused by burns.

Material and Methods Study design This was a pilot study. The protocol was approved by out institution's research ethics committee and registered in ClinicalTrials. The study adhered to the principles of the Declaration of Helsinki, and informed consent was obtained from all participants prior to enrollment. This was conducted in compliance with the TITAN Guidelines 2025 (11).

Participants All participants were admitted to the Department of Rehabilitation Medicine for the first time after complete epithelialization of the wound. Eligible inclusion criteria are defined as participants who underwent skin grafting after suffering from deep second- or third degree burns around the mouth, and who complained of difficulties in daily life such as difficulty in eating, pronunciation, and oral hygine care due to microstomia (Figure 1). Exclusion criteria included patients diagnosed with limited temporomandibular joint movement after or before burn injury, at risk of skin damage when wearing an open mouthpiece, with bleeding at the scar site or scar at risk of epidermal damage, with peripheral vascular diseases with reduced blood circulation, and who withdrew consent.

Manufacturing patient-tailored mouthpiece using 3D modeling technology Each participant's mouths were scanned using a 3D scanner (Peel 3, Peel 3D, Canada) with a mesh resolution of 0.25 mm to create the mouthpiece model. Optical 3D scanning took 15 minutes, including setup. The scanned model was exported in (STL file) format. The model was imported into the modeling software (Geomagic Design X, 3D Systems, USA), in which sculpt mode was selected for further processing. 'Mouthpiece' tool was then selected followed by manual highlighting of the area of interest which included the following zones; the longest horizontal and vertical length of the mouth, and lip thickness. Computer-aided design (CAD) was completed in approximately 2 hours by using CAD model creation software Geomagic Design X®. The resulting mouthpiece was exported as .STL file. The STL file was imported into PreForm software, oriented and support was generated, and the print job was sent to the 3D printer. The mouthpiece part was printed using a Stereo Lithography Apparatus(SLA) 3D printer (Form 4B Medical, Formlabs, USA) that uses a light source to cure liquid resin, and the material was a high-strength biocompatible photopolymer resin (BioMed Clear Resin) (12). 3D printing of the mouthpiece took approximately 1 hour and 30 minutes. The printed part was placed in a Formlabs-validated wash unit (Form Wash, Formlabs, USA) containing 99% isopropyl alcohol for 15 minutes or until clean. Remove the part from the wash unit and soak in fresh isopropyl alcohol for 5 minutes. Remove the part and let it air dry at room temperature for at least 30 minutes. Place the dried part in a Formlabs-validated post-curing unit (Form Cure, Formlabs, USA) and cure at 60°C for 60 minutes. After the support of the cured mouthpiece was removed with a part removal tool or by hand, and then sanded smooth with sandpaper to improve the surface finish (Figure 2).

Intervention The participant was advised to wear the appliance throughout the day except during meals. The maximaum horizontal and vertical distances were measured every two weeks to assess whether the mouthpiece had the ability to stretch against the scar. If the patient found it easy to wear or there was no stretching effect, the patient-tailored mouthpiece was remade.

All participants had the same daily schedule and performed their daily routine, including eating, showering, rehabilitation therapy, and scar management such as using moisturizing cream. Nonsurgical treatments such as intralesional steroid injection, moisturization, massage, silicone apply, and compression garment were maintained to suppress hypertrophic scars during the period of wearing the mouthpiece.

Outcome measurements A clinical researcher conducted a blind assessment of scar biological properties before applying the mouthpiece and after application. As a primary outcome, the vertical and horizontal lengths of the mouth were measured before and after wearing the patient-customized mouthpiece for 2 months. As defined previously in the article, vertical mouth opening range wea recorded as the measurement in millimeters from the inner border of the medial top lip to the inner border of the medial lower lip whilist in the stretched position. Horizontal mouth opening range was recorded as the measurement in millimeters from one lateral oral commissure to the other lateral oral commissure whilst in the stretched position (Figure 3) (13). As secondary outcomes, the biological scar properties, the Vancouver Scar Scale (VSS), and the Patient and Observer Scar Assessment Scale (POSAS) scores were evaluated before and after applying the mouthpiece for 2 months. The VSS was used to assess and evaluate scar severity. Scar evaluation involved individual assessment of four factors; pigmentation, vascularity, pliability, and scar height (thickness). Each parameter was scored on a scale from 0 to3 or 0 to 5, with 0 representing normal skin and higher scores indicating increased severity or deviation from normality. The total score was calculated by summing the individual scores for each parameter, providing an overall assessment of scar severity (14). The POSAS is a consistent and reliable tool designed to assess scars, particularly burn scars, from both the patient's and observer's perspectives. It consists of two numeric scale; one for patients, encompassing six parameters, and the other for observers, comprising five parameters (15).

The space for skin examination was maintained at 40~50% humidity and 20~25'C (16). Scar thickness was quantified using ultrasonography (128 BW1 US system, Medison, Korea) (8). The Mexameter® (MX18, Courage-Khazaka Electronics GmbH, Köln, Germany) was used to measure melanin levels and erythema severity. Higher values indicated greater pigmentation and redness. Trans-epidermal water loss (TEWL) was measured using a Tewameter® (Courage-Khazaka Electronic GmbH, Köln, Germany) to evaluate water evaporation. Possible complications, including pain, ecchymosis, skin abrasion, and swelling, were also monitored.

Statistical analysis Statistical analysis was performed using SPSS 23.0 (IBM Corporation, Armonk, NY, USA). Due to the small sample size, nonparametric methods were applied. The Wilcoxon signed-rank test was used for in-group comparisons of the variables. Statistical significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* who underwent skin grafting after suffering from deep second- or third degree burns around the mouth
* who complained of difficulties in daily life such as difficulty in eating, pronunciation, and oral hygine care due to microstomia

Exclusion Criteria:

* diagnosed with limited temporomandibular joint movement after or before burn injury
* at risk of skin damage when wearing an open mouthpiece
* with bleeding at the scar site or scar at risk of epidermal damage
* with peripheral vascular diseases with reduced blood circulation
* who withdrew consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
mouth size measurement | 2 month
  vertical mouth opening range wea recorded as the measurement in millimeters from the inner border of the medial top lip to the inner border of the medial lower lip whilist in the stretched position. Horizontal mouth opening range was recorded as the measurement in millimeters from one lateral oral commissure to the other lateral oral commissure whilst in the stretched position

SECONDARY OUTCOMES:
Vancouver Scar Scale (VSS) | 2 months
  The VSS was used to assess and evaluate scar severity. Scar evaluation involved individual assessment of four factors; pigmentation, vascularity, pliability, and scar height (thickness). Each parameter was scored on a scale from 0 to3 or 0 to 5, with 0 representing normal skin and higher scores indicating increased severity or deviation from normality. The total score was calculated by summing the individual scores for each parameter, providing an overall assessment of scar severity

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Scared Heart Hospital IRB, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Singounas EG. Posttraumatic brainstem damage. Surg Neurol. 1986 Sep;26(3):311. doi: 10.1016/0090-3019(86)90171-0. No abstract available. PMID 3738730
- [Result] Joo SY, Lee SY, Cho YS, Yi S, Seo CH. Clinical Utility of an Exoskeleton Robot Using Three-Dimensional Scanner Modeling in Burn Patient: A Case Report. J Burn Care Res. 2021 Sep 30;42(5):1030-1034. doi: 10.1093/jbcr/irab060. PMID 33881533
- [Result] Ki SH, Jo GY, Yoon J, Choi MSS. Reconstruction of microstomia considering their functional status. Arch Craniofac Surg. 2020 Jun;21(3):161-165. doi: 10.7181/acfs.2020.00220. Epub 2020 Jun 29. PMID 32630987